CLINICAL TRIAL: NCT04739449
Title: '4C' Intervention to Reduce SARS-CoV-2 Transmission: Coaching, Cleaning, Communication and Collaboration
Brief Title: '4C' Intervention to Reduce SARS-CoV-2 (Covid-19) Transmission
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Since the vaccine there are no COVID 19 cases in proposed study sites.
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lona Mody, Amanda Sanford Hickey Collegiate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00186126; 3P30AG024824-16S1 (NIH)
Record Dates: First submitted 2021-02-03; First posted 2021-02-04 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV Infection; Covid19
Keywords: Environmental Contamination; Nursing Home; Interventions
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: The study will have a cluster-randomized design in which two of the four nursing homes will be randomized to the intervention arm or the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Two facilities will follow their local protocols for infection prevention, including COVID-19 precautions. We will swab environmental surfaces at these sites to compare outcomes.
- Intervention (Experimental): Using a cluster-randomized design, we will test a multimodal aging-friendly intervention including four components (4Cs):
  1. Coaching staff
  2. Cleaning protocols, standardized
  3. Communication with staff and leadership
  4. Collaboration with local expertise
  We hypothesize that the implementation of this organizational QI educational program will be associated with lower odds of SARS-CoV-2 transmission to the environment.
  Interventions: Behavioral: Coaching, Cleaning, Communication, Collaboration

INTERVENTIONS:
Behavioral: Coaching, Cleaning, Communication, Collaboration — 1. Coaching staff
  2. Cleaning protocols, standardized
  3. Communication with staff and leadership
  4. Collaboration with local expertise
  Arms: Intervention

SUMMARY:
Nursing homes have long faced special challenges in implementing effective infection prevention programs, including limited resources and diagnostic challenges in a frail functionally disabled long-stay population. Advancing our understanding of the transmission of SARS-CoV-2 within these facilities for vulnerable populations deserves urgent and further investigation. Environmental contamination with SARS-CoV-2 that is reported in limited studies highlights the potential importance of transmission between patients, their environment, and healthcare providers via direct and indirect contact.

This study seeks to characterize the epidemiology of SARS-CoV- 2 in the NH patient room environment over time and the risk of transmission to near and far environments, with the explicit intent of developing integrated, simple COVID-19 infection prevention strategies that can be reported to and implemented throughout other nursing homes and long-term care facilities.

DETAILED DESCRIPTION:
In order to achieve these goals the study is being performed at four different nursing homes and will include patients with active or with recent COVID-19 infection, as well as nursing home staff members. The study will test a multimodal aging-friendly intervention including four components and hypothesizes that the implementation of this organizational, educational, quality improvement program will be associated with lower odds of SARS-CoV-2 transmission to the environment.

ELIGIBILITY:
Inclusion criteria for nursing home patients:

* 18 years of age or older
* Residing in a participating nursing home facility
* Active or recent (last 14 days) COVID-19 infection

Exclusion criteria for nursing home patients:

* Not located in a participating nursing home facility

Inclusion criteria for healthcare workers:

- Healthcare worker at a participating nursing home facility

Exclusion criteria for healthcare workers:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-04 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Surface contamination with SARS-CoV-2 | 3 months, depending on COVID-19 epidemiology
  Prevalence of SARS-CoV-2 on surfaces in COVID-19 positive patient rooms

IPD SHARING:
Plan to Share IPD: No